CLINICAL TRIAL: NCT06940284
Title: Food Intake of Hospitalized Elderly and Its Influence on Muscular and Clinical Outcomes: A Prospective Cohort Study
Brief Title: Food Intake of Hospitalized Elderly and Its Influence on Muscular and Clinical Outcomes
Status: Recruiting | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Hamilton Augusto Roschel da Silva, PhD, University of Sao Paulo General Hospital
Other Study IDs: 66834923300000068
Record Dates: First submitted 2025-04-14; First posted 2025-04-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Atrophy, Muscular; Undernutrition
MeSH Terms: conditions — Muscular Atrophy; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older individuals hospitalized: Older adults admitted to the hospital within the past 48 hours, without signs of delirium, and able to receive oral nutrition and complete muscle function assessments.

SUMMARY:
The objectives of the present study are: 1) to characterize the energy-protein intake of the elderly during hospitalization; 2) to verify the influence of energy-protein intake during hospitalization on muscular (i.e., cross-sectional area of the rectus femoris and vastus lateralis muscles, muscle strength, functionality and level of independence) and clinical (i.e., length of hospital stay, hospital readmission and mortality) at the time of hospital discharge, 2 and 6 months after hospital discharge and; 3) to verify whether energy-protein intake during hospitalization is a significant predictor of loss of function and muscle mass, length of hospital stay, hospital readmission rate and mortality.

ELIGIBILITY:
Inclusion Criteria:

* both sex;
* 65 years and older;
* hospital stay less than 48 hours;

Exclusion Criteria:

* cancer in the last 5 years;
* delirium;
* cognitive deficit that impossibility the patient to read and sign the informed consent form;
* neurological disease;
* neurodegenerative muscular disease;
* patients receive nutrition via enteral and parenteral routes.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older individuals hospitalized
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Vastus Lateralis Muscle Cross-sectional Area | From date of admission until the date of medical discharge. Up to 30 days.
  Vastus Lateralis Muscle Cross-sectional Area will be assessed through ultrasound

SECONDARY OUTCOMES:
Handgrip strength | From date of admission until the date of medical discharge. Up to 30 days.
  Strength will be evaluated using handgrip strength test
Muscle function | From date of admission until the date of medical discharge. Up to 30 days.
  Muscle function evaluated trough battery of test
Functional independence | From date of admission until the date of medical discharge. Up to 30 days.
  Functional independence will be assessed using Barthel Index. The scores range from 0 to 100. A score of 100 means the individual is fully independent, while lower scores indicate increasing levels of dependence.
Length of hospital stay | From date of admission until the date of medical discharge. Up to 30 days.
  Length of hospital stay will be the time (in days) until medical discharge.
Mortality | From date of admission until the date of medical discharge. Up to 30 days.
  Mortality rate in percent
Hospital readmission post-medical discharge | 1- and 2- months post-medical discharge
  Hospital readmission post-medical discharge will be the number of times that he is admitted in the hospital post-medical discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Hamilton Roschel, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No